CLINICAL TRIAL: NCT07333131
Title: Identification of Iatrogenic Drug Events Upon Admission to the Adult Emergency Departments
Acronym: IATRO-URG
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9542
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Iatrogenic Drug Events
Keywords: Iatrogenic drug events; Pharmaceutical intervention; Medication-related iatrogenesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pharmacists working within a multidisciplinary team have a role to play in detecting the potential iatrogenic origin of a hospital admission, in order to implement measures to improve medication use appropriately and limit readmissions for medication-related iatrogenesis. The iatrogenic detection process depends on the individual involved, their experience, and any tools consulted. Indeed, detection aids have their place in this process and aim for better identification. For example, a questionnaire called AT HARM 10 was developed by a team of experienced pharmacists to identify hospitalizations related to medication-related iatrogenesis. The use of this tool has been validated for pharmacists as well as for pharmacy students: interns and fifth-year medical students.

Identifying iatrogenic drug events among patients presenting to the emergency department using the AT HARM 10 grid in order to intervene and adapt therapeutic management. This clinical pharmacy activity complements what is already included in routine care (medication review, pharmaceutical analysis, and pharmaceutical intervention to adapt treatment).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (> 65 years old)
* Treated in the emergency department of Hautepierre Hospital
* Presenting a prioritization score > 7 according to the Von Korff score
* Subject (and their legal representative, if applicable) not objecting to the reuse of their data for scientific research purposes.

Exclusion Criteria:

- Presence of a written objection in the patient's medical file (and/or that of their legal representative, if applicable) to the reuse of their data for scientific research purposes

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adult patient (> 65 years old) treated in the emergency department of Hautepierre Hospital and presenting a prioritization score > 7 according to the Von Korff score
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients for whom an iatrogenic event was identified | Up to 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pharmacie - Stérilisation - CHU de Strasbourg - France, Strasbourg, France